CLINICAL TRIAL: NCT07081971
Title: Effect of the Bioheat Patch on Pain Following the HyFoSy Procedure
Acronym: B-HyP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Yaakov Melcer, Professor yaakov melcer, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0130-25-ASF
Record Dates: First submitted 2025-05-21; First posted 2025-07-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Pain; Infertility; Pain Management; Gynecologic Procedures
MeSH Terms: conditions — Pelvic Pain; Infertility; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: 40 women will receive the active Bioheat patch. (Experimental)
  Interventions: Other: Bioheat Patch
- Control Group: 40 women will receive a non-heating placebo patch (Experimental)
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Other: Bioheat Patch — Bioheat Patch for pain relif
  Arms: Intervention Group: 40 women will receive the active Bioheat patch.
Other: Placebo Patch — placebo Patch
  Arms: Control Group: 40 women will receive a non-heating placebo patch

SUMMARY:
This randomized controlled trial (RCT) evaluates the efficacy of Bioheat thermal patches in reducing post-procedural pain following Hysterosalpingo Foam Sonography (HyFoSy).

HyFoSy is a common ultrasound-based diagnostic procedure to assess tubal patency and uterine cavity structure in women undergoing fertility workup. While generally less painful than HSG, many patients still report moderate to severe cramping and discomfort during and after the test.

Thermal therapy has demonstrated effectiveness in reducing musculoskeletal and gynecological pain. Bioheat patches, approved by the Israeli Ministry of Health for menstrual pain relief, emit safe, low-grade heat (approximately 37-38°C) and may provide a non-invasive pain management strategy post-HyFoSy.

Participants (n=80) will be women aged 20-45 undergoing HyFoSy. They will be randomly assigned to either the Bioheat intervention group or a placebo patch group, applied externally to the lower abdomen. The heat-producing patch contains iron and other safe materials that react with oxygen to emit continuous heat without electricity. Infrared radiation from the patch components may also promote local vasodilation and muscle relaxation.

Pain assessment will use the validated Visual Analog Scale (VAS), collected post-procedure via follow-up SMS and phone contact. The study aims to quantify reduction in perceived pain, and potentially improve patient satisfaction with HyFoSy. Safety has been pre-established, with no reported adverse skin effects when used as instructed.

Study duration is six months, following ethics approval at the OB-GYN ultrasound department of Shamir Medical Center.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18-45 scheduled for HyFoSy

No dermatologic conditions at the patch site

No allergies to patch ingredients, or heat

No active pelvic infections

Exclusion Criteria:

Active genital infection

Skin issues in lower abdomen

Sensitivity to heat

Any medical condition preventing local heat use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by Visual Analog Scale (VAS) | Up to 6 hours post-procedure
  Pain will be assessed using the VAS (range: 0-10; 0 = no pain, 10 = worst imaginable pain). Participants will self-report their score via questionnaire within 6 hours after the procedure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melcer Y, Nimrodi M, Levinsohn-Tavor O, Gal-Kochav M, Pekar-Zlotin M, Maymon R. Analgesic Efficacy of Intrauterine Lidocaine Flushing in Hysterosalpingo-foam Sonography: A Double-blind Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Aug;28(8):1484-1489. doi: 10.1016/j.jmig.2020.11.019. Epub 2020 Nov 26. PMID 33249268